CLINICAL TRIAL: NCT06833255
Title: Thriving Beyond Breast Cancer: Post-Treatment Supportive Services Programming for Breast Cancer Survivors to Optimize Health During Survivorship
Brief Title: A Post-treatment Supportive Service Program for the Transition Into Survivorship for Black Women Breast Cancer Survivors in Western New York
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I-4133324; NCI-2024-10482 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4133324 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (survivorship support) (Experimental): Patients attend survivorship group support sessions over 2 hours on the 1st and 3rd Thursday of each month and 1:1 peer mentoring sessions with long-term breast cancer survivors on the 2nd and 4th Thursday of each month for up to 12 months.
  Interventions: Other: Interview; Other: Questionnaire Administration; Other: Support; Procedure: Support Group Therapy

INTERVENTIONS:
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Other: Support — Attend 1:1 peer mentoring sessions
  Other Names: Supportive - procedure intent
Procedure: Support Group Therapy — Attend survivorship group support sessions

SUMMARY:
This clinical trial studies whether a post-treatment supportive service program can be used to help breast cancer survivors in Western New York (WNY) transition into post-treatment life (survivorship). The post-treatment supportive service program is delivered to breast cancer survivors of WNY. It combines group support sessions and one-on-one (1:1) peer mentoring sessions. The group support sessions include traditional support groups, educational topics/lessons, activities, such as cooking lessons, celebrations, or facility tours, and guest speakers. The 1:1 peer mentoring sessions are held with a long-term breast cancer survivor mentor. The long-term breast cancer survivor mentor helps the mentee get in the practice of performing once monthly self-assessments and create plans to help improve any identified modifiable risk factors. The long-term breast cancer survivor mentor can also help connect the mentee to providers or resources as needed. A post-treatment supportive service program may help Black women breast cancer survivors in WNY transition into survivorship.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Design, develop, and deliver a no-cost, culturally appropriate, community-engaged, evidence-based, easily accessible, multilevel program to one hundred individuals who are breast cancer survivors in WNY prioritzing those who have most recently transitioned into their post-treatment life and/or self-identify as African American.

SECONDARY OBJECTIVES:

I. Determine the feasibility and acceptability of the newly generated survivorship programming.

II. Prepare for possible future dissemination and implementations at other National Witness Project® (NWP) sites.

EXPLORATORY OBJECTIVES:

I. Examinations of:

Ia. Program participants overall health, wellbeing, and quality of life; Ib. Program participants breast cancer recurrence rates; Ic. Factors that influence the program's self-sustainability potential; Id. Processes involved in programming revision / modification / improvement etc.

OUTLINE:

Patients attend survivorship group support sessions over 2 hours on the 1st and 3rd Thursday of each month and 1:1 peer mentoring sessions with long-term breast cancer survivors on the 2nd and 4th Thursday of each month for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and read English
* At least 18 years of age or older
* Live in the Western New York area
* Has been diagnosed with breast cancer (any stage)
* Has completed primary breast cancer treatments (i.e., systemic, radiation, and/or surgical interventions other than breast reconstruction surgeries)

  * Mentors are at least one-year post-treatment completion
  * Mentees are less than one-year post-treatment completion
  * Note: Individuals who have completed primary breast cancer treatments who are being managed with ongoing hormonal therapies and/or are awaiting breast reconstruction surgery may participate in this study (i.e., these therapies do not meet exclusion criteria)

    * Note: Although any breast cancer survivor may participate, priority will be given to those who have most recently transitioned into their post-treatment life (or those who report that support was either not offered or was unavailable to them during their less recent transition into post-treatment life) and /or self-identify as African American

Exclusion Criteria:

* Currently receiving neoadjuvant and/or adjuvant systemic and/or radiations therapies
* Unwilling or unable to complete the assessment in English
* Are pregnant or nursing
* Are unwilling or unable to follow protocol requirements

  * Note: Individuals who have completed primary breast cancer treatments who are being managed with ongoing hormonal therapies and/or are awaiting breast reconstruction surgery may participate in this study (i.e., these therapies do not meet exclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Community-clinical linkages | Up to 12 months
  Will assess the number of community-clinical linkages between organizations that support enrollment of breast cancer survivors who are Black into grant survivorship services. This will include formal agreements with at least: 1 cancer center, 2 primary care facilities, and 4 community organizations.
Facilitators to implementation | At 6 and 12 months
  Will be assessed using semi-structured interviews conducted at focus groups. An integrated (i.e., both deductive and inductive) approach to data analysis will be used. Qualitative data analyses techniques will be used to identify key themes within and across the interviewee groups. A structured summary template will be created using key elements from the interviewee guides to organize and condense data based on Consolidated Framework for Implementation Research (CFIR) domains. At least two implementation evaluation team members will participate in the initial coding of interviews and synthesis of summary sheets. Summary sheets will be transferred into matrix displays by the main coder (Devonish) and categorized into barriers and facilitators within each CFIR domain for each interviewee group. Group matrices will then be compared to determine cross-cutting themes and explore differences across groups.
Barriers to implementation | At 6 and 12 months
  Will be assessed using semi-structured interviews conducted at focus groups. An integrated (i.e., both deductive and inductive) approach to data analysis will be used. Qualitative data analyses techniques will be used to identify key themes within and across the interviewee groups. A structured summary template will be created using key elements from the interviewee guides to organize and condense data based on CFIR domains. At least two implementation evaluation team members will participate in the initial coding of interviews and synthesis of summary sheets. Summary sheets will be transferred into matrix displays by the main coder (Devonish) and categorized into barriers and facilitators within each CFIR domain for each interviewee group. Group matrices will then be compared to determine cross-cutting themes and explore differences across groups.

SECONDARY OUTCOMES:
Enrollment rate | Up to 12 months
  Will be assessed using very basic mathematical equations, no advanced level statistical analyses will be involved.
Retention rate | Up to 12 months
  Will be assessed using very basic mathematical equations, no advanced level statistical analyses will be involved.
Acceptability of intervention | Up to 12 months
  Feedback will be compiled into a quarterly summary report that will be distributed during the execution phase of the proposed programming. Quarterly reports will be available for board members' quarterly meetings during the execution phase to guide shared decision making about content changes, adjustments, and guest facilitators.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Devonish, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States